CLINICAL TRIAL: NCT02649829
Title: First-line Immunotherapy Using Wilms' Tumor Protein 1 (WT1)-Targeted Dendritic Cell Vaccinations for Malignant Pleural Mesothelioma
Brief Title: Autologous Dendritic Cell Vaccination in Mesothelioma
Acronym: MESODEC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other); Stichting tegen Kanker (Other)
Responsible Party: Principal Investigator, Zwi Berneman, Study coordinator, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRG13-002
Record Dates: First submitted 2015-12-07; First posted 2016-01-08 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: dendritic cell vaccination; chemo-immunotherapy; Wilms' tumor 1 (WT1)
MeSH Terms: conditions — Mesothelioma, Malignant; Wilms Tumor | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): dendritic cell vaccination plus chemotherapy
  Interventions: Biological: dendritic cell vaccination plus chemotherapy

INTERVENTIONS:
Biological: dendritic cell vaccination plus chemotherapy — A. Chemoimmunotherapy:
  1. four 3-weekly cycles of platinum/pemetrexed; on day 1 of each cycle, pemetrexed 500 mg/m2 should be administered as intravenous (IV) infusion over 10 minutes followed 30 minutes later by cisplatin 75 mg/m2 as IV over approximately 2 hours.
  2. four intradermal vaccinations with 8-10 x 10e6 autologous WT1 mRNA-loaded DCs; at day 14+/- 3 days after the start of each chemotherapy cycle.
  B. Surgery: pleurectomy/decortication; in case of resectable disease, 4-6 weeks after start of the last chemotherapy cycle.
  Other Names: chemoimmunotherapy

SUMMARY:
In this multicenter phase I/II trial, dendritic cells (DCs) loaded with the mesothelioma-associated tumor antigen WT1 will be used in conjunction with conventional chemotherapy for the frontline treatment of malignant pleural mesothelioma (MPM). The general objective is to provide the first-in-human experimental demonstration that the combination of platinum/pemetrexed-based chemotherapy with WT1-targeted DC vaccination is feasible and safe and enables the induction of both systemic and in situ mesothelioma-specific immune responses in patients with MPM.

DETAILED DESCRIPTION:
Malignant pleural mesothelioma (MPM) is a highly aggressive and in virtually all cases fatal cancer that is tightly associated with prior asbestos exposure. Despite some improvement over time, the prognosis of patient diagnosed with MPM remains dismal with a median overall survival from diagnosis of only 12 months.

In this single arm phase I/II trial the investigators want to demonstrate the feasibility and safety of WT1-targeted dendritic cell vaccination in MPM patients as frontline treatment in conjunction with first line platinum/pemetrexed-based chemotherapy and the induction of both systemic and in situ mesothelioma-specific immune responses. During three years of recruitment the investigators aim at including 20 patients diagnosed with histologically proven epithelial MPM (WHO grade 0-1) who are able to undergo leukapheresis, chemotherapy, immunotherapy and pleurectomy/decortication (P/D; in case of resectable disease). Patients who underwent prior treatment for MPM or with a history of another malignancy within the last five years will be excluded.

The intention of this study is to administer four vaccine doses in combination with standard of care of four 3-weekly cytoreductive platinum/pemetrexed-based chemotherapy cycles to each participant and prior to surgery (P/D) in the case of resectable MPM. Patients will receive four 3-weekly intradermal vaccinations with autologous WT1 messenger (m)RNA-loaded dendritic cells (V1-4), at day 14 after the start of each chemotherapy cycle (CT1-4).

The dendritic cell therapy product will be generated and administered in the Antwerp University Hospital, more specifically the Center for Cell Therapy and Regenerative Medicine (CCRG) and the Division of Hematology, both headed by Prof. Zwi Berneman.

The DC vaccines will be under embargo from release until the safety and quality control test results have become available and all release criteria have been met. A detailed overview of all applicable release criteria is provided in the investigational medicinal product dossier. The embargo period generally lasts 3 weeks counting from the day of cryopreservation (i.e. 8 days after leukapheresis).

Recruitment started in August 2017. Study-related follow-up of the included patients is intended to be until 90 days after final DC vaccine administration or 22 months after diagnosis, whichever occurs later. In addition to feasibility and safety of the chemoimmunotherapy schedule, the investigators will look for the time to progression (TTP), progression-free survival (PFS), overall survival (OS), systemic immunogenicity and local immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis with histologically proven epithelial
* Aged ≥ 18 years at the time of enrollment
* WHO performance status 0-1 at the time of enrollment
* Fit to undergo general anesthesia, a thoracoscopy, leukapheresis, chemotherapy, immunotherapy and P/D (in case of resectable disease)
* No history of receiving any investigational treatment within 28 days of study enrollment
* No history of intolerance to pemetrexed and/or cisplatin
* Women of child bearing potential must have negative serum or urine pregnancy test at the time of screening. They should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least hundred days after the last study treatment. If pregnancy does occur within this time period, the Principal investigator must be informed as soon as possible. Female subjects who are breastfeeding should discontinue nursing prior to the first dose of study treatment and until hundred days after the last study treatment
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discusses with the patient before registration in the trial. Absence of any other inability or unwillingness to comply with the requirements of the protocol as assessed by the investigator
* Before patient registration written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Unwilling or unable to comply with the study requirements
* Prior treatment for MPM
* History of another malignancy within the last five years (except for carcinoma in situ of the cervix, basal cell or spinocellular carcinoma of the skin or unless the investigator rationalizes otherwise)
* Known proven metastases
* Known concomitant presence of any immunosuppressive disease (e.g. HIV) or any active autoimmune condition, except for vitiligo
* Pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
Number of MPM patients with feasible and safe DC vaccine production | Vaccine production and quality testing (i.e. 4 weeks after leukapheresis)
  Production of autologous DC vaccines from newly diagnosed MPM patients will be evaluated for:
  1. Feasibility, assessed by success of leukapheresis and production of sufficient (i.e. at least 4 vaccines) and qualified (phenotypic and functional requirements) vaccines.
  2. Safety, assessed by microbiological testing (bacteria, yeast, fungi, mycoplasma, endotoxin) of the DC vaccines.
Number of patients receiving investigational DC vaccine administration combined with standard of care chemotherapy within the proposed time frame | After the chemoimmunotherapy treatment (+/- 15 weeks after entry to trial)
  Administration of 4 autologous DC vaccines combined with four 3-weekly platinum/pemetrexed-based chemotherapy cycles will be evaluated for:
  1. Feasibility, assessed by successful administration of DC vaccines and prior to surgery in case of resectable disease.
  2. Safety, assessed by local (e.g. skin reactions at injection site) and systemic (toxicity grading according to the latest version of the CTCAE and CTC ) tolerability to the treatment.

SECONDARY OUTCOMES:
Objective clinical responses by tumor evaluation (clinical efficacy) | Through study completion, at least after 4 DC vaccinations, prior to surgery (in case of resectable disease) + three months after the last intervention and within every 12 months during follow-up
  Objective clinical responses to the chemoimmunotherapy and, in case of resectable disease, after surgery as compared to baseline tumor evaluation prior to treatment (i.e. at diagnosis), will be evaluated with:
  1. radiographic assessments (CT imaging) of the tumor response using the modified RECIST criteria.
  2. FDG-PET assessments of the tumor response using the PERCIST criteria.
  Patients will be followed for disease progression; time to progression (TTP) and progression-free survival (PFS).
Overall survival (clinical efficacy) | Through study completion, an average of 1 year
  Patients will be followed for survival, from diagnosis and from start of treatment, for which the accurate date and reason of death (cancer-related or non-related) will be recorded for every patient.
Systemic immunogenicity | After the fourth DC vaccine (i.e. post chemoimmunotherapy, prior to surgery in case of resectable disease)
  Systemic immunogenicity will be evaluated by:
  1. Detection of WT1-specific T cell immunity and innate immunity in peripheral blood.
  2. Response to delayed-type hypersensitivity (DTH) skin testing to the DC vaccine.
Local immunogenicity | Upon surgery (P/D)
  Local immunogenicity will be evaluated by detection of immune profile in tumor biopsies and/or pleurectomy specimens (in case of resectable disease).

CONTACTS AND LOCATIONS:
Overall Officials: Zwi N Berneman, MD, PhD, Study Director — Antwerp University Hospital, Division of Hematology and Center for Cell Therapy and Regenerative Medicine; Eva Lion, MSc, PhD, Principal Investigator — University of Antwerp, Laboratory of Experimental Hematology; Evelien LJ Smits, MSc, PhD, Principal Investigator — University of Antwerp, Laboratory of Experimental Hematology; Sébastien Anguille, MD, PhD, Principal Investigator — Antwerp University Hospital, Division of Hematology
Locations (3):
- Belgium (3):
  - Antwerp University Hospital, Edegem, Antwerp
  - AZ Middelares, Ghent
  - AZ Nikolaas, Sint-Niklaas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robinson BW, Musk AW, Lake RA. Malignant mesothelioma. Lancet. 2005 Jul 30-Aug 5;366(9483):397-408. doi: 10.1016/S0140-6736(05)67025-0. PMID 16054941
- [Background] Robinson BW, Lake RA. Advances in malignant mesothelioma. N Engl J Med. 2005 Oct 13;353(15):1591-603. doi: 10.1056/NEJMra050152. No abstract available. PMID 16221782
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Musk AW, Olsen N, Alfonso H, Reid A, Mina R, Franklin P, Sleith J, Hammond N, Threlfall T, Shilkin KB, de Klerk NH. Predicting survival in malignant mesothelioma. Eur Respir J. 2011 Dec;38(6):1420-4. doi: 10.1183/09031936.00000811. Epub 2011 Jul 7. PMID 21737558
- [Background] Bagia M, Nowak AK. Novel targeted therapies and vaccination strategies for mesothelioma. Curr Treat Options Oncol. 2011 Jun;12(2):149-62. doi: 10.1007/s11864-011-0149-1. PMID 21424750
- [Background] Bograd AJ, Suzuki K, Vertes E, Colovos C, Morales EA, Sadelain M, Adusumilli PS. Immune responses and immunotherapeutic interventions in malignant pleural mesothelioma. Cancer Immunol Immunother. 2011 Nov;60(11):1509-27. doi: 10.1007/s00262-011-1103-6. Epub 2011 Sep 13. PMID 21913025
- [Background] Izzi V, Masuelli L, Tresoldi I, Foti C, Modesti A, Bei R. Immunity and malignant mesothelioma: from mesothelial cell damage to tumor development and immune response-based therapies. Cancer Lett. 2012 Sep 1;322(1):18-34. doi: 10.1016/j.canlet.2012.02.034. Epub 2012 Mar 3. PMID 22394996
- [Background] Gregoire M. What's the place of immunotherapy in malignant mesothelioma treatments? Cell Adh Migr. 2010 Jan-Mar;4(1):153-61. doi: 10.4161/cam.4.1.11361. Epub 2010 Jan 30. PMID 20179421
- [Background] Kushitani K, Takeshima Y, Amatya VJ, Furonaka O, Sakatani A, Inai K. Immunohistochemical marker panels for distinguishing between epithelioid mesothelioma and lung adenocarcinoma. Pathol Int. 2007 Apr;57(4):190-9. doi: 10.1111/j.1440-1827.2007.02080.x. PMID 17316414
- [Background] Anguille S, Smits EL, Lion E, van Tendeloo VF, Berneman ZN. Clinical use of dendritic cells for cancer therapy. Lancet Oncol. 2014 Jun;15(7):e257-67. doi: 10.1016/S1470-2045(13)70585-0. PMID 24872109
- [Background] Hegmans JP, Hemmes A, Aerts JG, Hoogsteden HC, Lambrecht BN. Immunotherapy of murine malignant mesothelioma using tumor lysate-pulsed dendritic cells. Am J Respir Crit Care Med. 2005 May 15;171(10):1168-77. doi: 10.1164/rccm.200501-057OC. Epub 2005 Mar 11. PMID 15764728
- [Background] Hegmans JP, Veltman JD, Lambers ME, de Vries IJ, Figdor CG, Hendriks RW, Hoogsteden HC, Lambrecht BN, Aerts JG. Consolidative dendritic cell-based immunotherapy elicits cytotoxicity against malignant mesothelioma. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1383-90. doi: 10.1164/rccm.200909-1465OC. Epub 2010 Feb 18. PMID 20167848
- [Background] Smits EL, Anguille S, Cools N, Berneman ZN, Van Tendeloo VF. Dendritic cell-based cancer gene therapy. Hum Gene Ther. 2009 Oct;20(10):1106-18. doi: 10.1089/hum.2009.145. PMID 19656053
- [Background] Van Tendeloo VF, Ponsaerts P, Lardon F, Nijs G, Lenjou M, Van Broeckhoven C, Van Bockstaele DR, Berneman ZN. Highly efficient gene delivery by mRNA electroporation in human hematopoietic cells: superiority to lipofection and passive pulsing of mRNA and to electroporation of plasmid cDNA for tumor antigen loading of dendritic cells. Blood. 2001 Jul 1;98(1):49-56. doi: 10.1182/blood.v98.1.49. PMID 11418462
- [Background] Van Tendeloo VF, Van de Velde A, Van Driessche A, Cools N, Anguille S, Ladell K, Gostick E, Vermeulen K, Pieters K, Nijs G, Stein B, Smits EL, Schroyens WA, Gadisseur AP, Vrelust I, Jorens PG, Goossens H, de Vries IJ, Price DA, Oji Y, Oka Y, Sugiyama H, Berneman ZN. Induction of complete and molecular remissions in acute myeloid leukemia by Wilms' tumor 1 antigen-targeted dendritic cell vaccination. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13824-9. doi: 10.1073/pnas.1008051107. Epub 2010 Jul 14. PMID 20631300
- [Background] Benteyn D, Anguille S, Van Lint S, Heirman C, Van Nuffel AM, Corthals J, Ochsenreither S, Waelput W, Van Beneden K, Breckpot K, Van Tendeloo V, Thielemans K, Bonehill A. Design of an Optimized Wilms' Tumor 1 (WT1) mRNA Construct for Enhanced WT1 Expression and Improved Immunogenicity In Vitro and In Vivo. Mol Ther Nucleic Acids. 2013 Nov 19;2(11):e134. doi: 10.1038/mtna.2013.54. PMID 24253259
- [Background] Treasure T, Lang-Lazdunski L, Waller D, Bliss JM, Tan C, Entwisle J, Snee M, O'Brien M, Thomas G, Senan S, O'Byrne K, Kilburn LS, Spicer J, Landau D, Edwards J, Coombes G, Darlison L, Peto J; MARS trialists. Extra-pleural pneumonectomy versus no extra-pleural pneumonectomy for patients with malignant pleural mesothelioma: clinical outcomes of the Mesothelioma and Radical Surgery (MARS) randomised feasibility study. Lancet Oncol. 2011 Aug;12(8):763-72. doi: 10.1016/S1470-2045(11)70149-8. Epub 2011 Jun 30. PMID 21723781
- [Background] Lang-Lazdunski L, Bille A, Lal R, Cane P, McLean E, Landau D, Steele J, Spicer J. Pleurectomy/decortication is superior to extrapleural pneumonectomy in the multimodality management of patients with malignant pleural mesothelioma. J Thorac Oncol. 2012 Apr;7(4):737-43. doi: 10.1097/JTO.0b013e31824ab6c5. PMID 22425923
- [Background] McCoy MJ, Nowak AK, Lake RA. Chemoimmunotherapy: an emerging strategy for the treatment of malignant mesothelioma. Tissue Antigens. 2009 Jul;74(1):1-10. doi: 10.1111/j.1399-0039.2009.01275.x. Epub 2009 May 4. PMID 19422663
- [Background] Galluzzi L, Senovilla L, Zitvogel L, Kroemer G. The secret ally: immunostimulation by anticancer drugs. Nat Rev Drug Discov. 2012 Feb 3;11(3):215-33. doi: 10.1038/nrd3626. PMID 22301798
- [Background] Park S, Schalling M, Bernard A, Maheswaran S, Shipley GC, Roberts D, Fletcher J, Shipman R, Rheinwald J, Demetri G, et al. The Wilms tumour gene WT1 is expressed in murine mesoderm-derived tissues and mutated in a human mesothelioma. Nat Genet. 1993 Aug;4(4):415-20. doi: 10.1038/ng0893-415. PMID 8401592
- [Background] Cheever MA, Allison JP, Ferris AS, Finn OJ, Hastings BM, Hecht TT, Mellman I, Prindiville SA, Viner JL, Weiner LM, Matrisian LM. The prioritization of cancer antigens: a national cancer institute pilot project for the acceleration of translational research. Clin Cancer Res. 2009 Sep 1;15(17):5323-37. doi: 10.1158/1078-0432.CCR-09-0737. PMID 19723653
- [Background] Krug LM, Dao T, Brown AB, Maslak P, Travis W, Bekele S, Korontsvit T, Zakhaleva V, Wolchok J, Yuan J, Li H, Tyson L, Scheinberg DA. WT1 peptide vaccinations induce CD4 and CD8 T cell immune responses in patients with mesothelioma and non-small cell lung cancer. Cancer Immunol Immunother. 2010 Oct;59(10):1467-79. doi: 10.1007/s00262-010-0871-8. Epub 2010 Jun 8. PMID 20532500
- [Background] Van Driessche A, Berneman ZN, Van Tendeloo VF. Active specific immunotherapy targeting the Wilms' tumor protein 1 (WT1) for patients with hematological malignancies and solid tumors: lessons from early clinical trials. Oncologist. 2012;17(2):250-9. doi: 10.1634/theoncologist.2011-0240. Epub 2012 Jan 30. PMID 22291091
- [Background] Hsu FJ, Benike C, Fagnoni F, Liles TM, Czerwinski D, Taidi B, Engleman EG, Levy R. Vaccination of patients with B-cell lymphoma using autologous antigen-pulsed dendritic cells. Nat Med. 1996 Jan;2(1):52-8. doi: 10.1038/nm0196-52. PMID 8564842
- [Background] Wahl RL, Jacene H, Kasamon Y, Lodge MA. From RECIST to PERCIST: Evolving Considerations for PET response criteria in solid tumors. J Nucl Med. 2009 May;50 Suppl 1(Suppl 1):122S-50S. doi: 10.2967/jnumed.108.057307. PMID 19403881
- [Background] Hoos A. Evolution of end points for cancer immunotherapy trials. Ann Oncol. 2012 Sep;23 Suppl 8:viii47-52. doi: 10.1093/annonc/mds263. PMID 22918928
- [Background] Anguille S, Smits EL, Bryant C, Van Acker HH, Goossens H, Lion E, Fromm PD, Hart DN, Van Tendeloo VF, Berneman ZN. Dendritic Cells as Pharmacological Tools for Cancer Immunotherapy. Pharmacol Rev. 2015 Oct;67(4):731-53. doi: 10.1124/pr.114.009456. PMID 26240218
- [Background] Qi XW, Zhang F, Wu H, Liu JL, Zong BG, Xu C, Jiang J. Wilms' tumor 1 (WT1) expression and prognosis in solid cancer patients: a systematic review and meta-analysis. Sci Rep. 2015 Mar 9;5:8924. doi: 10.1038/srep08924. PMID 25748047
- [Background] Thomas A, Chen Y, Yu T, Gill A, Prasad V. Distinctive clinical characteristics of malignant mesothelioma in young patients. Oncotarget. 2015 Jun 30;6(18):16766-73. doi: 10.18632/oncotarget.4414. PMID 26202904
- [Background] Panou V, Vyberg M, Weinreich UM, Meristoudis C, Falkmer UG, Roe OD. The established and future biomarkers of malignant pleural mesothelioma. Cancer Treat Rev. 2015 Jun;41(6):486-95. doi: 10.1016/j.ctrv.2015.05.001. Epub 2015 May 8. PMID 25979846
- [Background] Nowak AK, Cook AM, McDonnell AM, Millward MJ, Creaney J, Francis RJ, Hasani A, Segal A, Musk AW, Turlach BA, McCoy MJ, Robinson BW, Lake RA. A phase 1b clinical trial of the CD40-activating antibody CP-870,893 in combination with cisplatin and pemetrexed in malignant pleural mesothelioma. Ann Oncol. 2015 Dec;26(12):2483-90. doi: 10.1093/annonc/mdv387. Epub 2015 Sep 18. PMID 26386124
- [Background] Marcq E, Pauwels P, van Meerbeeck JP, Smits EL. Targeting immune checkpoints: New opportunity for mesothelioma treatment? Cancer Treat Rev. 2015 Dec;41(10):914-24. doi: 10.1016/j.ctrv.2015.09.006. Epub 2015 Sep 28. PMID 26433514
- [Background] Fisher SA, Cleaver A, Lakhiani DD, Khong A, Connor T, Wylie B, Lesterhuis WJ, Robinson BW, Lake RA. Neoadjuvant anti-tumor vaccination prior to surgery enhances survival. J Transl Med. 2014 Sep 4;12:245. doi: 10.1186/s12967-014-0245-7. PMID 25186961
- [Background] Berneman ZN, Van de Velde AL, Willemen Y, Anguille S, Saevels K, Germonpré P, Huizing MT, Peeters M, Snoeckx A, Parizel P, Van Tendeloo VF, Lion E, Nijs G, Stein B, Vermeulen K, Maes MB, Malfait R, Vrelust I, Verlinden A, Gadisseur AP, Schroyens WA, Lammens M and Smits EL. Blood 124(21): 310-310, 2014.
- [Background] Berneman Z, Germonpre P, Huizing MT, Van De Velde A, Nijs G, Stein B, Van Tendeloo V, Lion E, Smits EL and Anguille S. J Clin Oncol 32:5s(suppl): abstr 7583, 2014.
- [Background] Adusumilli PS. Translational immunotherapeutics: chemoimmunotherapy for malignant pleural mesothelioma. Cancer. 2014 Nov 1;120(21):3268-71. doi: 10.1002/cncr.28883. Epub 2014 Jul 2. No abstract available. PMID 24989696
- [Background] Coosemans A, Vanderstraeten A, Tuyaerts S, Verschuere T, Moerman P, Berneman ZN, Vergote I, Amant F, VAN Gool SW. Wilms' Tumor Gene 1 (WT1)--loaded dendritic cell immunotherapy in patients with uterine tumors: a phase I/II clinical trial. Anticancer Res. 2013 Dec;33(12):5495-500. PMID 24324087
- [Background] Coosemans A, Vanderstraeten A, Tuyaerts S, Verschuere T, Moerman P, Berneman Z, Vergote I, Amant F, Van Gool SW. Immunological response after WT1 mRNA-loaded dendritic cell immunotherapy in ovarian carcinoma and carcinosarcoma. Anticancer Res. 2013 Sep;33(9):3855-9. PMID 24023319
- [Background] Willemen Y, Huizing MT, Smits E, Anguille S, Nijs G, Stein B, Van Tendeloo V, Peeters M, Berneman Z. J Clin Oncol 30(suppl): abstr e13051, 2012.
- [Background] Anguille S, Van de Velde AL, Smits EL, Van Tendeloo VF, Juliusson G, Cools N, Nijs G, Stein B, Lion E, Van Driessche A, Vandenbosch I, Verlinden A, Gadisseur AP, Schroyens WA, Muylle L, Vermeulen K, Maes MB, Deiteren K, Malfait R, Gostick E, Lammens M, Couttenye MM, Jorens P, Goossens H, Price DA, Ladell K, Oka Y, Fujiki F, Oji Y, Sugiyama H, Berneman ZN. Dendritic cell vaccination as postremission treatment to prevent or delay relapse in acute myeloid leukemia. Blood. 2017 Oct 12;130(15):1713-1721. doi: 10.1182/blood-2017-04-780155. Epub 2017 Aug 22. PMID 28830889
- [Background] Z. Berneman, A. Van de Velde, S. Anguille, Y. Willemen, M. Huizing, P. Germonpré, K. Saevels, G. Nijs, N. Cools, A. Van Driessche, B. Stein, H. De Reu, W. Schroyens, A. Gadisseur, A. Verlinden, K. Vermeulen, M. Maes, M. Lammens, H. Goossens, M. Peeters, V. Van Tendeloo, E. Smits. Vaccination with Wilms' Tumor Antigen (WT1) mRNA-Electroporated Dendritic Cells as an Adjuvant Treatment in 60 Cancer Patients: Report of Clinical Effects and Increased Survival in Acute Myeloid Leukemia, Metastatic Breast Cancer, Glioblastoma and Mesothelioma. Cytotherapy 2016, 18(6), p. S13-14
- [Background] Z. Berneman, S. Anguille, Y. Willemen, A. Van de Velde, P. Germonpré, M. Huizing, V. Van Tendeloo, K. Saevels, L. Rutsaert, K. Vermeulen, A. Snoeckx, B. Op de Beeck, N. Cools, G. Nijs, B. Stein, E. Lion, A. van Driessche, M. Peeters, E. Smits. Vaccination of cancer patients with dendritic cells electroporated with mRNA encoding the Wilms' Tumor protein (WT1): correlation of clinical effect and overall survival with T-cell response. Cytotherapy 2019, 21(5), p. S10.